CLINICAL TRIAL: NCT00258323
Title: A Phase II Trial of Pre- and Postoperative Chemoradiotherapy and ZD1839 (IRESSA) Followed by Maintenance ZD1839 in Patients With Locoregionally Advanced Esophageal and Gastroesophageal Junction Carcinoma
Brief Title: Radiotherapy,Chemotherapy,Before and After Surgery in Advanced Esophageal or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCF5848; P30CA043703 (NIH); CCF-5848 (Other: Cleveland Clinic IRB); ZENECA-1839/US/0233
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Fluorouracil; Gefitinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin — 20mg/m2d/IV continuous infusion x days
  Other Names: CDDP
Drug: fluorouracil — 1000mg/m2/d IV continuous infusion x 4 days
  Other Names: 5 FU
Drug: Iressa — 250mg po qd days 1-28 then x 2 years
  Other Names: ZD 1839
Procedure: conventional surgery — conventional surgery
Radiation: radiation therapy — 150 cGy bid

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Cisplatin and fluorouracil may also make tumor cells more sensitive to radiation therapy. Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving radiation therapy together with combination therapy and gefitinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving radiation therapy together with combination chemotherapy and gefitinib before and after surgery works in treating patients with advanced esophageal or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the activity of gefitinib, in terms of median survival and distant metastatic disease control, in patients treated with neoadjuvant and adjuvant cisplatin, fluorouracil, and radiotherapy who are undergoing surgery for esophageal and gastroesophageal junction cancer.

Secondary

* Determine the pathologic complete and partial response rate in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients and in patients who are disease free and receiving long-term maintenance gefitinib.

OUTLINE:

* Preoperative regimen: Patients undergo radiotherapy twice a day during days 1-12 (for a total of 10 treatment days). Patients receive fluorouracil IV continuously and cisplatin IV continuously on days 1-4. Patients also receive oral gefitinib once daily on days 1-28. At 6 weeks, patients with locoregionally confined disease undergo surgical resection and then proceed to the postoperative regimen. Patients with a medical contraindication to surgery proceed directly to the postoperative regimen.
* Postoperative regimen: Beginning 4-10 weeks after surgery or 6 weeks after completing the first course of therapy, patients undergo radiotherapy and receive fluorouracil and cisplatin as in the preoperative regimen.
* Maintenance regimen: Patients receive oral gefitinib beginning on day 1 of the postoperative regimen and continuing for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma, adenocarcinoma, or large cell undifferentiated cancer of the esophagus or gastroesophageal junction

  * T3, N1, or M1a disease only
  * The following types are not allowed:

    * Small cell undifferentiated carcinomas, lymphomas, or sarcomas
    * Small cell or mixed small cell/non-small cell histology
* No evidence of distant hematogenous tumor metastases (M1b)
* No malignant pleural effusions

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC > 3,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Alkaline phosphatase < 2 times normal
* AST < 2 times normal
* No unstable or uncompensated hepatic disease

Renal

* Creatinine ≤ 2.0 mg/dL
* Calcium normal
* No unstable or uncompensated renal disease

Cardiovascular

* No unstable or uncontrolled angina
* No unstable or uncompensated cardiac disease

Pulmonary

* See Disease Characteristics
* No limitations to pulmonary function that would preclude study participation
* No evidence of clinically active interstitial lung disease (asymptomatic patients with chronic stable radiographic changes are allowed)
* No unstable or uncompensated respiratory disease

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No evidence of severe or uncontrolled systemic disease
* No other uncontrolled malignancy
* No active infection
* No known severe hypersensitivity to gefitinib or any of its excipients

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for this cancer

Chemotherapy

* No prior chemotherapy for this cancer

Radiotherapy

* No prior radiotherapy for this cancer

Surgery

* Recovered from any prior oncologic or other major surgery
* No prior surgical resection for this cancer
* No concurrent ophthalmic surgery

Other

* No prior photodynamic therapy for this cancer (prior laser treatments are acceptable)
* More than 30 days since prior unapproved or investigational drug
* No concurrent phenytoin, carbamazepine, barbiturates, rifampin, phenobarbital, or Hypericum perforatum (St. John's wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-10; Primary Completion 2007-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Survival at 1 year | 1 year
  Survival at 1 year
Distant metastatic control at 1 year | 1 year
  Distant metastatic control at 1 year

SECONDARY OUTCOMES:
Response rate at 6 weeks | 6 weeks
  Response rate at 6 weeks
Toxicity of induction chemoradiotherapy and gefitinib as measured by CTC version 2.0 at 6 weeks | 6 weeks
  Toxicity of induction chemoradiotherapy and gefitinib as measured by CTC version 2.0 at 6 weeks
Toxicity of maintenance gefitinib as measured by CTC version 2.0 every 8 weeks after the completion of radiotherapy | 8 weeks
  Toxicity of maintenance gefitinib as measured by CTC version 2.0

CONTACTS AND LOCATIONS:
Overall Officials: David J. Adelstein, MD, Study Chair — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/results?term=ccf5848